CLINICAL TRIAL: NCT07124741
Title: Prognostic Power of the VEXUS Score in Septic Shock: Efficacy in Mortality Prediction
Brief Title: Prognostic Power of the VEXUS Score in Septic Shock: Effectiveness in Mortality Prediction
Status: Not yet recruiting | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nilgun Kavrut Ozturk, Professor, Antalya Training and Research Hospital
Other Study IDs: 2024-435
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Septic Shock; VExUS
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic shock cohort: All patients diagnosed with septic shock in the ıntensive care unit will undergo serial ultrasonographic evaluations to calculate the VEXUS Score at 0-4 hours, 12-24 hours, and 72 hours. These scores will be analyzed in relation to 28-day mortality. No treatment decisions will be made based on the VEXUS results.
  Interventions: Diagnostic Test: Serial VEXUS Ultrasound Evaluation

INTERVENTIONS:
Diagnostic Test: Serial VEXUS Ultrasound Evaluation — Ultrasound assessments will be performed by an experienced anesthesiologist at three time points (0-4 hours, 12-24 hours, and 72 hours)to determine the degree of venous congestion using the VEXUS Score. No treatment changes will be made based on the VEXUS findings. The scores will solely be used for prognostic correlation with mortality outcomes.

SUMMARY:
This study aims to evaluate the prognostic power of the VEXUS Score in predicting mortality among patients with septic shock in intensive care units.

DETAILED DESCRIPTION:
After the diagnosis of septic shock, patients will be assessed for eligibility. Following informed consent, measurements will be taken within the first 4 hours of shock onset, and treatment (inotropic and vasopressor doses, fluid challenge, corticosteroids) will be recorded. A second measurement will occur between 12 and 24 hours, and a third at 72 hours. All treatment and care protocols will be managed according to routine unit protocols.

Data will be systematically collected at three time points (0-4 hours, 12-24 hours, and 72 hours). These will include hemodynamic parameters, laboratory tests (including infection markers), need for renal replacement therapy, mechanical ventilation requirement and duration, cumulative dose and duration of vasopressor use, ICU stay, and survival status.

VEXUS Score Grading

The VEXUS score will be graded as follows:

* Grade 0 (No Congestion): No signs of venous congestion are detected. The inferior vena cava (IVC) diameter is less than 2 cm.
* Grade 1 (Mild Venous Congestion): The IVC diameter is 2 cm or greater. However, hepatic, portal, or renal vein flow measurements exhibit normal waveform patterns, or only one mildly abnormal waveform pattern is present.
* Grade 2 (Moderate Venous Congestion): The IVC diameter is 2 cm or greater. Additionally, analysis of hepatic, portal, or renal vein waveforms reveals one severe congestion finding.
* Grade 3 (Severe Venous Congestion): The IVC diameter is 2 cm or greater. Furthermore, analysis of hepatic, portal, or renal vein waveforms shows two or more severe congestion findings.

Data will be analyzed using SPSS version 23.0, with normality assessed through visual and analytical methods (Kolmogorov-Smirnov/Shapiro-Wilk tests). Continuous variables will be compared using t-tests or Mann-Whitney U tests, and categorical variables using Chi-square tests. ROC analysis will be used to assess the predictive value of VEXUS for mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Patients monitored for septic shock in intensive care unit
* Signed informed consent

Exclusion Criteria:

* Age <18
* Severe obesity precluding adequate ultrasonographic imaging.
* Patients in whom venous structures cannot be clearly assessed via ultrasonography due to anatomical or technical reasons (e.g., adhesions following abdominal surgery).
* Patients receiving dialysis due to chronic kidney disease or initiating dialysis for acute kidney failure.
* Chronic heart failure.
* Patients with advanced valvular insufficiency or advanced pulmonary hypertension.
* Patients with portal hypertension or advanced-stage liver cirrhosis.
* Presence of acute or chronic thrombosis in the inferior vena cava or other venous structures within the scoring area.
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the intensive care unit with a diagnosis of septic shock according to Sepsis-3 criteria. Patients will be enrolled consecutively from the intensive care unit of a tertiary care university hospital. Informed consent will be obtained from all patients or their legal representatives.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
28-day intensive care unit mortality in relation to VEXUS score | Up to 28 days following intensive care unit admission.
  Investigation of the relationship between VEXUS Score and 28-day mortality in patients diagnosed with septic shock in the intensive care unit.

SECONDARY OUTCOMES:
Need for mechanical ventilation in relation to VEXUS score | Within the first 72 hours of intensive care unit admission.
  Evaluation of the association between initial VEXUS score and the requirement for mechanical ventilation in patients
Duration of mechanical ventilation in relation to VEXUS score. | From intensive care unit patients admission until extubation, up to 28 days.
  Assessment of the correlation between VEXUS scores and the total duration of mechanical ventilation in intensive care unit patients with septic shock.
Length of intensive care unit stay in relation to VEXUS score | From intensive care unit admission until intensive care unit discharge, up to 28 days.
  Investigation of the association between VEXUS score pregression and total length of intensive care unit stay in patients with septic shock.
Vasopressor dose and duration in relation to VEXUS score. | First 72 hours after intensive care unit admission
  Assessment of the relationship between serial VEXUS scores and the cumulative dose and duration of vasopressor therapy during the first 72 hours in patients diagnosed with septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Kavrut Ozturk, Professor, Study Chair — University of Health Sciences Antalya Training and Research hospital